CLINICAL TRIAL: NCT04026776
Title: Uric Acid, Klotho and Salt Sensitivity in Young Adults Born Preterm
Acronym: PEPC3
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00057527; 1R01HL146818-01A1 (NIH)
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-04

CONDITIONS: Salt; Excess; Blood Pressure Disorders
Keywords: Uric Acid sensitivity; Salt sensitivity; Blood Pressure Influences
MeSH Terms: interventions — Allopurinol; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preterm Group (Experimental): Subjects with very low birth weight (<37 completed weeks' gestation and birth weight <1500 g) will receive a dietary intervention (high/low salt diet) and FDA approved drug, Allopurinol
  Interventions: Drug: Allopurinol; Other: Dietary Intervention
- Term-born control group (Active Comparator): Subjects with birth weight ≥2500 g will receive a dietary intervention (high/low salt diet)
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Drug: Allopurinol — Study Part 2- Preterm group only: After Visit 5 preterm born participants will start allopurinol 200 mg daily PO for 6 weeks. The 1 week high and low salt diets and assessments will be repeated while on allopurinol.
  Other Names: Zyloprim
  Arms: Preterm Group
Other: Dietary Intervention — High-Na+ (250 mmol/d) and low-Na+ (50 mmol/d) standard isocaloric K+ diets (75 mmol/1000 kcal/d) for 1 week each as 3 meals and 1 snack a day provided by the Clinical Research Unit Metabolic Kitchen. Part 2 preterm only- the diets will be repeated while the participant is taking allopurinol.

SUMMARY:
The purpose of this research is to learn about how salt in the diet influences blood pressure in young adults who were born prematurely.

DETAILED DESCRIPTION:
Premature birth is an emerging and important risk factor for hypertension and cardiovascular disease, as both preterm birth rates and infant survival increase worldwide. Hypertension and cardiovascular disease begin in early adulthood in individuals born prematurely, but the reasons especially in regard to the role of preterm birth are unknown. An improved understanding of why hypertension and cardiovascular disease occur in early adulthood in individuals born preterm will enable the development of prevention and treatment strategies to mitigate the burden of cardiovascular disease. Investigators propose to investigate these relationships mechanistically in a clinical trial of subjects born preterm to establish the SSBP (salt sensitivity of blood pressure) phenotype and study its relationship to CVD (cardiovascular disease) compared to a control group of healthy term- born peers. Investigators will then propose to determine if blocking UA (uric acid) formation improves SSBP and cardiovascular function in subjects born preterm.

ELIGIBILITY:
Inclusion Criteria:

* Singleton birth
* Born at less than 34 weeks gestational age (preterm cohort)
* Born at greater than 36 weeks gestational age (term cohort)

Exclusion Criteria:

* Twin birth
* Congenital anomalies or genetic syndromes
* Currently pregnant or breast feeding
* Subject-reported history of hypertension
* Current use of antihypertensive medications
* Active cancer
* Chronic kidney disease
* Heart failure
* Liver failure

Ages: 22 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proportion with salt sensitivity of blood pressure at baseline via ABPM | Day 7 to 14
  Defined as a ≥8 mmHg decrease in mean arterial blood pressure when moving from the high-Na+ to the low-Na+ phase, as measured on 24-hour ambulatory blood pressure monitoring (ABPM).
Proportion with salt sensitivity of blood pressure after allopurinol via ABPM | Day 49 to 56
  A ≥8 mmHg decrease in mean arterial blood pressure when moving from the high-Na+ to the low-Na+ phase while taking allopurinol, as measured on 24-hour ambulatory blood pressure monitoring (ABPM).
Salt sensitivity index at baseline | Day 7 to 14
  The ratio between the change in 24-hour mean arterial pressure, as measured on 24-hour ambulatory blood pressure monitoring, and the change in 24-hour urine Na+ concentration when moving from the high-Na+ phase to the low-Na+ phase.
Salt sensitivity index after allopurinol | Day 49 to 56
  The ratio between the change in 24-hour mean arterial pressure, as measured on 24-hour ambulatory blood pressure monitoring, and the change in 24-hour urine Na+ concentration when moving from the high-Na+ phase to the low-Na+ phase while taking allopurinol
Proportion with salt sensitivity of blood pressure at baseline via casual blood pressure | Day 7 to 14
  A >=5 mmHg decrease in mean arterial blood pressure measured in clinic when moving from the high-Na+ phase to the low-Na+ phase. Casual blood pressure measured 3 consecutive times via auscultation with the average of the 3 mean arterial blood pressure measurements recorded.
Proportion with salt sensitivity of blood pressure after allopurinol via casual blood pressure | Day 49 to 56
  A >=5 mmHg decrease in mean arterial blood pressure measured in clinic when moving from the high-Na+ phase to the low-Na+ phase while taking allopurinol. Casual blood pressure measured 3 consecutive times via auscultation with the average of the 3 mean arterial blood pressure measurements recorded.
High blood pressure at baseline via ABPM | Day 0
  Proportion with 24-hour mean systolic or diastolic blood pressure ≥115/75 mmHg, awake mean systolic or diastolic blood pressure ≥120/80 mmHg, or asleep mean systolic or diastolic blood pressure ≥100/65 mmHg, measured with ambulatory blood pressure monitoring (ABPM).
Hypertension at baseline via ABPM | Day 7
  Proportion with 24-hour mean systolic or diastolic blood pressure ≥125/75 mmHg, awake mean systolic or diastolic blood pressure ≥130/80 mmHg, or asleep mean systolic or diastolic blood pressure ≥110/65 mmHg, measured with ambulatory blood pressure monitoring (ABPM).
High blood pressure at baseline via casual blood pressure | First 3 study visits
  Proportion with mean systolic or diastolic blood pressure ≥120/80 mmHg, measured via 3 consecutive auscultated measurements (averaged) at each of 3 separate study visits.
Hypertension at baseline via casual blood pressure | First 3 study visits
  Proportion with mean systolic or diastolic blood pressure ≥130/80 mmHg, measured via 3 consecutive auscultated measurements (averaged) at each of 3 separate study visits
Serum uric acid at baseline | Day 0
  Serum uric acid concentration at baseline
Change in serum uric acid with dietary Na+ intervention | Day 7 to 14
  The change in serum uric acid levels when moving from high-Na+ phase to the low-Na+ phase
Change in serum uric acid with dietary Na+ intervention on allopurinol | Day 42 to 56
  The change in serum uric acid levels when moving from high-Na+ phase to the low-Na+ phase while on allopurinol
Pulse wave velocity at baseline | Day 0
  Carotid femoral pulse wave velocity will be measured at baseline with the SphygmoCor XCEL device
Augmentation index at baseline | Day 0
  Augmentation index will be measured at baseline with the SphygmoCor XCEL device
Heart rate variability at baseline | Day 0
  Heart rate variability will be measured at baseline using continuous heart rate recording using the CNAP™ Monitor 500i
Baroreflex sensitivity at baseline | Day 0
  Baroreflex sensitivity will be measured at baseline using continuous blood pressure and heart rate using the CNAP™ Monitor 500i
Angiotensin-(1-7) at baseline | Day 0
  Plasma angiotensin-(1-7) concentration and urine angiotensin-(1-7)/creatinine at baseline
Angiotensin II at baseline | Day 0
  Plasma angiotensin II concentration and urine angiotensin II/creatinine at baseline
Klotho at baseline | Day 0
  Plasma klotho concentration and urine klotho/creatinine at baseline.
Creatinine at baseline | Day 0
  Serum creatinine concentration at baseline
Cystatin C at baseline | Day 0
  Serum cystatin C concentration at baseline
eGFR at baseline | Day 0
  Estimated glomerular filtration rate (eGFR) at baseline.We will calculate the eGFR by the CKD-EPI Creatinine-Cystatin C 2012 equation and by 24 hour creatinine

SECONDARY OUTCOMES:
Ambulatory systolic blood pressure 24-hour mean at baseline | Day 0
  Average systolic blood pressure over 24 hours, measured with ambulatory blood pressure monitors
Ambulatory diastolic blood pressure 24-hour mean at baseline | Day 0
  Average diastolic blood pressure over 24 hours, measured with ambulatory blood pressure monitors
Ambulatory mean arterial pressure 24-hour mean at baseline | Day 0
  Average mean arterial pressure over 24 hours, measured with ambulatory blood pressure monitors
Ambulatory systolic blood pressure awake mean at baseline | Day 0
  Average systolic blood pressure while awake, measured with ambulatory blood pressure monitors
Ambulatory diastolic blood pressure awake mean at baseline | Day 0
  Average diastolic blood pressure while awake, measured with ambulatory blood pressure monitors
Ambulatory mean arterial pressure awake mean at baseline | Day 0
  Average mean arterial pressure while awake, measured with ambulatory blood pressure monitors
Ambulatory systolic blood pressure asleep mean at baseline | Day 0
  Average systolic blood pressure while asleep, measured with ambulatory blood pressure monitors
Ambulatory diastolic blood pressure asleep mean at baseline | Day 0
  Average diastolic blood pressure while asleep, measured with ambulatory blood pressure monitors
Ambulatory mean arterial pressure asleep mean at baseline | Day 0
  Average mean arterial pressure while asleep, measured with ambulatory blood pressure monitors
Ambulatory systolic blood pressure 24-hour load at baseline | Day 0
  Proportion of mean 24-hour systolic blood pressures ≥125 mmHg, measured with ambulatory blood pressure monitors
Ambulatory diastolic blood pressure 24-hour load at baseline | Day 0
  Proportion of mean 24-hour diastolic blood pressures ≥75 mmHg, measured with ambulatory blood pressure monitors.
Ambulatory systolic blood pressure awake load at baseline | Day 0
  Proportion of mean awake systolic blood pressures ≥130 mmHg, measured with ambulatory blood pressure monitors
Ambulatory diastolic blood pressure awake load at baseline | Day 0
  Proportion of mean awake diastolic blood pressures ≥80 mmHg, measured with ambulatory blood pressure monitors
Ambulatory systolic blood pressure asleep load at baseline | Day 0
  Proportion of mean asleep systolic blood pressures ≥110 mmHg, measured with ambulatory blood pressure monitors
Ambulatory diastolic blood pressure asleep load at baseline | Day 0
  Proportion of mean asleep diastolic blood pressures ≥65 mmHg, measured with ambulatory blood pressure monitors
Ambulatory systolic blood pressure nocturnal dipping at baseline | Day 0
  Percent change in mean awake to mean asleep systolic blood pressure, measured with ambulatory blood pressure monitors
Ambulatory diastolic blood pressure nocturnal dipping at baseline | Day 0
  Percent change in mean awake to mean asleep diastolic blood pressure, measured with ambulatory blood pressure monitors
Casual systolic blood pressure at baseline | Day 0
  Measured 3 consecutive times via auscultation with the average of the 3 systolic blood pressure measurements recorded
Casual diastolic blood pressure at baseline | Day 0
  Measured 3 consecutive times via auscultation with the average of the 3 diastolic blood pressure measurements recorded
Change in pulse wave velocity with dietary Na+ intervention | Day 7 to 14
  The change in carotid femoral pulse wave velocity will be measured with the SphygmoCor XCEL device when moving from high-Na+ phase to the low-Na+ phase
Change in augmentation index with dietary Na+ intervention | Day 7 to 14
  The change in augmentation index will be measured with the SphygmoCor XCEL device when moving from high-Na+ phase to the low-Na+ phase
Change in pulse wave velocity with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in carotid femoral pulse wave velocity will be measured with the SphygmoCor XCEL device when moving from high-Na+ phase to the low-Na+ phase while on allopurinol.
Change in augmentation index with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in augmentation index will be measured with the SphygmoCor XCEL device when moving from high-Na+ phase to the low-Na+ phase while on allopurinol
Change in heart rate variability with dietary Na+ intervention | Day 7 to 14
  The change in heart rate variability will be measured using the Continuous noninvasive arterial pressure (CNAP™) Monitor 500i when moving from high-Na+ phase to the low-Na+ phase
Change in baroreflex sensitivity with dietary Na+ intervention | Day 7 to 14
  The change in baroreflex sensitivity will be measured using the CNAP™ Monitor 500i when moving from high-Na+ phase to the low-Na+ phase
Change in heart rate variability with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in heart rate variability will be measured using the CNAP™ Monitor 500i when moving from high-Na+ phase to the low-Na+ phase while on allopurinol
Change in baroreflex sensitivity with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in baroreflex sensitivity will be measured using the CNAP™ Monitor 500i when moving from high-Na+ phase to the low-Na+ phase while on allopurinol
Change in angiotensin-(1-7) with dietary Na+ intervention | Day 7 to 14
  The change in plasma angiotensin-(1-7) concentration and urine angiotensin-(1-7)/creatinine when moving from the high-Na+ phase to the low-Na+ phase
Change in angiotensin II with dietary Na+ intervention | Day 7 to 14
  The change in plasma angiotensin II concentration and urine angiotensin II/creatinine when moving from the high-Na+ phase to the low-Na+ phase
Change in klotho with dietary Na+ intervention | Day 7 to 14
  The change in plasma klotho concentration and urine klotho/creatinine when moving from the high-Na+ phase to the low-Na+ phase
Change in angiotensin-(1-7) with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in plasma angiotensin-(1-7) concentration and urine angiotensin-(1-7)/creatinine when moving from the high-Na+ phase to the low-Na+ phase while on allopurinol
Change in angiotensin II with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in plasma angiotensin II concentration and urine angiotensin II/creatinine when moving from the high-Na+ phase to the low-Na+ phase while on allopurinol
Change in klotho with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in plasma klotho concentration and urine klotho/creatinine when moving from the high-Na+ phase to the low-Na+ phase while on allopurinol
ACE2 at baseline | Day 0
  Serum ACE2 concentration and activity and urine ACE2/creatinine and activity at baseline
ACE at baseline | Day 0
  Serum ACE concentration and activity and urine ACE/creatinine and activity at baseline
FGF23 at baseline | Day 0
  Plasma fibroblast growth factor 23 (FGF23) concentration and urine FGF23/creatinine at baseline
Change in ACE2 with dietary Na+ intervention | Day 7 to 14
  The change in serum ACE2 concentration and activity and urine ACE2/creatinine and activity when moving from the high-Na+ phase to the low-Na+ phase
Change in ACE2 with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in serum ACE2 concentration and activity and urine ACE2/creatinine and activity when moving from the high-Na+ phase to the low-Na+ phase while on allopurinol
Change in ACE with dietary Na+ intervention | Day 7 to 14
  The change in serum ACE concentration and activity and urine ACE2/creatinine and activity when moving from the high-Na+ phase to the low-Na+ phase
Change in ACE with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in serum ACE concentration and activity and urine ACE2/creatinine and activity when moving from the high-Na+ phase to the low-Na+ phase while on allopurinol
Change in FGF23 with dietary Na+ intervention | Day 7 to 14
  The change in serum fibroblast growth factor 23 (FGF23) concentration and urine FGF23/creatinine when moving from the high-Na+ phase to the low-Na+ phase
Change in FGF23 with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in serum fibroblast growth factor 23 (FGF23) concentration and urine FGF23/creatinine when moving from the high-Na+ phase to the low-Na+ phase while on allopurinol
Neprilysin level at baseline | Day 0
  Serum neprilysin concentration and activity and urine neprilysin/creatinine and activity at baseline
Change in neprilysin with dietary Na+ intervention | Day 7 to 14
  The change in serum neprilysin concentration and activity and urine neprilysin/creatinine and activity when moving from the high-Na+ phase to the low-Na+ phase
Change in neprilysin with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in serum neprilysin concentration and activity and urine neprilysin/creatinine and activity when moving from the high-Na+ phase to the low-Na+ phase while on allopurinol
Urine albumin at baseline | Day 0
  Urine albumin/creatinine at baseline on first-morning urine sample
Proportion with albuminuria | Day 0
  Albuminuria at baseline, defined as urine albumin/creatinine >30 mg/g on first-morning urine sample
Urine protein at baseline | Day 0
  Urine protein/creatinine at baseline on first-morning urine sample
Proportion with proteinuria | Day 0
  Proteinuria at baseline, defined as urine protein/creatinine >0.2 mg/mg on first-morning urine sample
Angiotensinogen at baseline | Day 0
  Serum angiotensinogen concentration and urine angiotensinogen/creatinine at baseline
Change in angiotensinogen with dietary Na+ intervention | Day 7 to 14
  The change in serum angiotensinogen concentration and urine angiotensinogen/creatinine when moving from the high-Na+ phase to the low-Na+ phase
Change in angiotensinogen with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in serum angiotensinogen concentration and urine angiotensinogen/creatinine when moving from the high-Na+ phase to the low-Na+ phase while on allopurinol
24-hour sodium excretion at baseline | Day 0
  Sodium excretion in the urine over 24 hours at baseline
24-hour potassium excretion at baseline | Day 0
  Potassium excretion in the urine over 24 hours at baseline
24-hour uric acid excretion at baseline | Day 0
  Uric acid excretion in the urine over 24 hours at baseline
Pulse wave velocity (CF) at baseline | Day 0
  Carotid-femoral (CF) pulse wave velocity will be measured at baseline with the SphygmoCor XCEL device
Change in pulse wave velocity (CF) with dietary Na+ intervention | Day 7 to 14
  The change in carotid-femoral (CF) pulse wave velocity will be measured with the SphygmoCor XCEL device when moving from high-Na+ phase to the low-Na+ phase
Change in pulse wave velocity (CF) with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in carotid-femoral (CF) pulse wave velocity will be measured with the SphygmoCor XCEL device when moving from high-Na+ phase to the low-Na+ phase while on allopurinol
Angiotensin II:angiotensin-(1-7) at baseline | Day 0
  Plasma and urine angiotensin II:angiotensin-(1-7) at baseline
Change in angiotensin II:angiotensin-(1-7) with dietary Na+ intervention | Day 7 to 14
  The change in plasma angiotensin II:angiotensin-(1-7) when moving from the high-Na+ phase to the low-Na+ phase
Change in angiotensin II:angiotensin-(1-7) with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in plasma angiotensin II:angiotensin-(1-7) when moving from the high-Na+ phase to the low-Na+ phase while on allopurinol
ACE:ACE2 at baseline | Day 0
  Serum and urine ACE:ACE2 at baseline
Change in ACE:ACE2 with dietary Na+ intervention | Day 7 to 14
  The change in serum and urine ACE:ACE2 when moving from the high-Na+ phase to the low-Na+ phase
Change in ACE:ACE2 with dietary Na+ intervention while on allopurinol | Day 49 to 56
  The change in serum and urine ACE:ACE2 when moving from the high-Na+ phase to the low-Na+ phase while on allopurinol
Body mass index at baseline | Day 0
  Body mass index at baseline
Proportion with overweight/obesity | Day 0
  Overweight/obesity at baseline, defined as a body mass index >=25 kg/m2
Proportion with obesity | Day 0
  Obesity at baseline, defined as a body mass index >=30 kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Shaltout, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results reported in this record, after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following publication.
Access Criteria: Proposals should be directed to hshaltou@wakehealth.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years.